CLINICAL TRIAL: NCT01950741
Title: An Single Arm, Single Dose Study to Evaluate the Effect of Intravitreal Injection of VEGF-Trap Eye on Polypoidal Choroidal Vasculopathy
Brief Title: Effect of Intravitreal VEGF-Trap Eye on Polypoidal Choroidal Vasculopathy
Acronym: VAULT
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Pusan National University Hospital (Other)
Collaborators: Bayer (Industry)
Responsible Party: Principal Investigator, Ji Eun Lee, Associate professor, Pusan National University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: D-1304-013-014
Record Dates: First submitted 2013-09-23; First posted 2013-09-25 (Estimated); Results first posted 2016-04-29 (Estimated); Last update posted 2016-04-29 (Estimated); Status verified 2016-03

CONDITIONS: Exudative Age-related Macular Degeneration; Polypoidal Choroidal Vasculopathy
MeSH Terms: conditions — Polypoidal Choroidal Vasculopathy | interventions — aflibercept

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- aflibercept (Experimental): Aflibercept 2 mg is injected into the vitreous cavity. Injections are given monthly three times, then are given bi-monthly to 12 months (month 0, 1, 2, 4, 6, 8, and 10; total 7 injections for 1 year).
  Interventions: Drug: aflibercept

INTERVENTIONS:
Drug: aflibercept — Aflibercept is injected intravitreally though the pars plana using 30G needle-attached syringe.
  Other Names: Eyelea, VEGF Trap-Eye

SUMMARY:
Effects of VEGF Trap-Eye (aflibercept) in treatment-naive polypoidal choroidal vasculopathy (PCV) will be evaluated.

DETAILED DESCRIPTION:
Efficacy of VEGF Trap-Eye (aflibercept, Eylea) for exudative age-related macular degeneration (AMD) was demonstrated in the phase III VIEW study. Polypoidal choroidal vasculopathy (PCV) is considered as a subtype of exudative AMD, however it is reportedly different from choroidal new vessels based on the histologic studies. The aim of this study is to evaluate effects of VEGF Trap-Eye in treatment of PCV, which was diagnosed using indocyanine green (ICG) angiography. VEGF Trap-Eye will be injected intravitreally bimonthly after 3 monthly loading dose for 12 months in treatment-naive PCV patients. The efficacy will be evaluated on preserving visual acuity and improving angiographic features at 12 months.

ELIGIBILITY:
Inclusion Criteria:

* Submacular PCV diagnosed using ICG angiography with no previous treatment (branching vascular network with or without polypoidal dilation in ICG angiography)
* Presence of signs of recent activity of PCV

  1. Visual acuity between 20/40 and 20/320
  2. Active leakage in fluorescein angiography
  3. Presence of any fluid in OCT(optical coherence tomography)-intraretinal, subretinal, sub-retinal pigment epithelial

Exclusion Criteria:

1. Extramacular PCV
2. Subretinal hemorrhage or other retinal lesions blocking angiographic characteristics in more than 50% area of PCV lesion.
3. Previous treatment of intravitreal injections (anti-VEGF, steroid or other agents)
4. Previous treatment of photodynamic therapy
5. Previous ocular surgery except cataract surgery before 3 or more months
6. Presence of exudative AMD in the other eyes requiring anti-VEGF treatment (Intravitreal bevacizumab was reported to affect the other eye.)
7. Presence of other ocular diseases which may affect visual acuity (glaucoma, cataract with opacity involving visual axis, etc)
8. Presence of uncontrolled systemic disease (diabetes mellitus, hypertension, ischemic heart disease, cerebral infarction, etc)
9. Patients who cannot understand or conform to the study protocol.
10. Patients who refuse to agree to the informed consent.
11. Patients with contraindication to aflibercept

    * Ocular or periocular infection
    * Active severe intraocular inflammation
    * Known hypersensitivity to aflibercept or to any of the excipients

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2013-09; Primary Completion 2015-05 (Actual); Study Completion 2015-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jae Pil Shin, MD, PhD, Study Director — Kyungbuk National University Hospital
Locations (8):
- South Korea (8):
  - Busan Paik Hospital, Busanjin-gu, Busan
  - Haeundae Paik Hospital, Haeundae, Busan
  - Gospel Hospital, Seo-gu, Busan
  - Pusan National University Hospital, Seo-gu, Busan
  - Keimyung University Dongsan Medical Center, Jung-gu, Daegu
  - Kyungpook National University Hospital, Jung-gu, Daegu
  - Yeungnam University Medical Center, Nam-gu, Daegu
  - Gyeongsang National University Hospital, Jinju, Gyeongsangnam-do

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Brown DM, Kaiser PK, Michels M, Soubrane G, Heier JS, Kim RY, Sy JP, Schneider S; ANCHOR Study Group. Ranibizumab versus verteporfin for neovascular age-related macular degeneration. N Engl J Med. 2006 Oct 5;355(14):1432-44. doi: 10.1056/NEJMoa062655. PMID 17021319
- [Background] Rosenfeld PJ, Brown DM, Heier JS, Boyer DS, Kaiser PK, Chung CY, Kim RY; MARINA Study Group. Ranibizumab for neovascular age-related macular degeneration. N Engl J Med. 2006 Oct 5;355(14):1419-31. doi: 10.1056/NEJMoa054481. PMID 17021318
- [Background] Heier JS, Brown DM, Chong V, Korobelnik JF, Kaiser PK, Nguyen QD, Kirchhof B, Ho A, Ogura Y, Yancopoulos GD, Stahl N, Vitti R, Berliner AJ, Soo Y, Anderesi M, Groetzbach G, Sommerauer B, Sandbrink R, Simader C, Schmidt-Erfurth U; VIEW 1 and VIEW 2 Study Groups. Intravitreal aflibercept (VEGF trap-eye) in wet age-related macular degeneration. Ophthalmology. 2012 Dec;119(12):2537-48. doi: 10.1016/j.ophtha.2012.09.006. Epub 2012 Oct 17. PMID 23084240
- [Background] Stangos AN, Gandhi JS, Nair-Sahni J, Heimann H, Pournaras CJ, Harding SP. Polypoidal choroidal vasculopathy masquerading as neovascular age-related macular degeneration refractory to ranibizumab. Am J Ophthalmol. 2010 Nov;150(5):666-73. doi: 10.1016/j.ajo.2010.05.035. Epub 2010 Aug 16. PMID 20719300
- [Background] Koh A, Lee WK, Chen LJ, Chen SJ, Hashad Y, Kim H, Lai TY, Pilz S, Ruamviboonsuk P, Tokaji E, Weisberger A, Lim TH. EVEREST study: efficacy and safety of verteporfin photodynamic therapy in combination with ranibizumab or alone versus ranibizumab monotherapy in patients with symptomatic macular polypoidal choroidal vasculopathy. Retina. 2012 Sep;32(8):1453-64. doi: 10.1097/IAE.0b013e31824f91e8. PMID 22426346

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Aflibercept
Started | 48
Completed | 45
Not Completed | 3
Not completed — Lost to Follow-up | 1
Not completed — Death | 1
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Arm/Group | Aflibercept
Number analyzed (Participants) | 48
Age, Continuous [Mean (Full Range); unit: years] | 68.3 [44 to 84]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 31
  Male | 17
Visual acuity [Mean (Standard Deviation); unit: letters] — Visual acuity was assessed using the Early Treatment Diabetic Retinopathy Study (ETDRS) chart. The ETDRS chart includes 100 letters as the maximum possible score, and 0 letters read as the minimum possible score. Higher scores represents better functioning. ETDRS letters of 85 are equivalent to 20/20 of vision.
  letters | 54.4 (18.1)

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Patients Lose Visual Acuity Less Than 15 Letters
Description: Visual acuity was assessed using the Early Treatment Diabetic Retinopathy Study (ETDRS) chart. The ETDRS chart includes 100 letters as the maximum possible score, and 0 letters read as the minimum possible score. Visual acuity of 85 letters is equivalent to 20/20. Higher scores represents better functioning.
Time Frame: 12 months
Population: Among 45 patients who completed the study, data of 5 were inadequate for the analysis. Forty patients were included in the analysis as per protocol set.
Measure: Number; unit: percentage of patients
Arm/Group | Aflibercept
Number analyzed (Participants) | 40
percentage of patients | 87.5

2. Secondary Outcome: Change in Visual Acuity From Baseline to 12 Months
Description: Mean changes of visual acuity in ETDRS letters. Visual acuity was assessed using ETDRS chart. The ETDRS chart includes 100 letters as the maximum possible score, and 0 letters read as the minimum possible score. Higher scores represents better functioning. A change of 5 letters is equivalent to a 1-line change.
Time Frame: Baseline and 12 months
Population: as for outcome 1
Measure: Mean (Full Range); unit: letters
Arm/Group | Aflibercept
Number analyzed (Participants) | 40
letters | 9 [-33 to 37]

3. Secondary Outcome: Percentage of Patients With Visual Acuity >=20/200
Description: Visual acuity was assessed using ETDRS chart. The ETDRS chart includes 100 letters as the maximum possible score, and 0 letters read as the minimum possible score. Higher scores represents better functioning. Percentage of patients with visual acuity 35 ETDRS letters (equivalent to 20/200) or better was calculated.
Time Frame: 12 months
Population: as for outcome 1
Measure: Number; unit: percentage of patients
Arm/Group | Aflibercept
Number analyzed (Participants) | 40
percentage of patients | 95.0

4. Secondary Outcome: Percentage of Patients With Visual Acuity >=20/40
Description: Visual acuity was assessed using ETDRS chart. The ETDRS chart includes 100 letters as the maximum possible score, and 0 letters read as the minimum possible score. Higher scores represents better functioning. Percentage of patients with visual acuity 70 ETDRS letters (equivalent to 20/40) or better was calculated.
Time Frame: 12 months
Population: as for outcome 1
Measure: Number; unit: percentage of patients
Arm/Group | Aflibercept
Number analyzed (Participants) | 40
percentage of patients | 52.5

5. Secondary Outcome: Percentage of Patients Having Complete Resulution of Polypoidal Lesion in ICG Angiography
Description: ICG angiography was assessed at 12 months. when no polypoidal lesion was detected, it was defined as complete resolution.
Time Frame: 12 months
Population: Among 45 patients who completed the study, data of 6 were inadequate for the analysis. 39 patients were included in the analysis.
Measure: Number; unit: percentage of patients
Arm/Group | Aflibercept
Number analyzed (Participants) | 39
percentage of patients | 66.7

6. Secondary Outcome: VFQ (Visual Function Questionaire)-25 Score
Description: Quality of life was assessed using VFQ -25 score . The VFQ-25 includes 25 questions, and the total score ranges from 0 to 100. Higher scores represents better functioning.
Time Frame: 12 months
Population: as for outcome 1
Measure: Mean (Inter-Quartile Range); unit: scores on a scale
Arm/Group | Aflibercept
Number analyzed (Participants) | 40
scores on a scale | 72.6 [67 to 77]

ADVERSE EVENTS:
Time Frame: Adverse events data was collected during the study perioid, or 1 year.
Groups:
- Aflibercept: Aflibercept 2 mg is injected into the vitreous cavity. Injections are given monthly three times, then are given bi-monthly to 12 months (month 0, 1, 2, 4, 6, 8, and 10; total 7 injections for 1 year).
  aflibercept: Aflibercept is injected intravitreally though the pars plana using 30G needle-attached syringe.
  Among 48 patients enrolled, one patient withdrew the consent before undergoing the first injection. Therefore the adverse event was assessed in 47 patients.
Arm/Group | Aflibercept
Serious Adverse Events (participants affected / at risk) | 1/47
Other Adverse Events (participants affected / at risk) | 4/47
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Aflibercept (N=47)
Death (Respiratory, thoracic and mediastinal disorders) | 1 (1) — Death resulted from pneumonia.
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Aflibercept (N=47)
Conjunctival hemorrhage (Eye disorders) | 4 (11)

LIMITATIONS AND CAVEATS:
Conjunctival hemorrhage is assessed based on medical records, and the incidence might be underestimated.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No